CLINICAL TRIAL: NCT06144931
Title: The Impact of Pericapsular Nerve Group Block on The Duration of Post-Operative Analgesia Following Hip Joint Surgeries
Brief Title: Efficacy of Pericapsular Nerve Group (PENG) Block for Hip Surgeries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Aiman Ahmad Al-Touny, Lecturer of Anesthesia and Intensive Care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4972#
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative
Keywords: PENG; Hip Joint Surgeries; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Patients in this group will be operated under spinal anesthesia
- PENG Group (Active Comparator): Patients in this group will undergo PENG block guided by ultrasound then spinal anesthesia will performed
  Interventions: Procedure: PENG Block

INTERVENTIONS:
Procedure: PENG Block — With the patient in the supine position, the ultrasound probe is placed on a transverse plane over the anterior superior iliac spine (ASIS). Once the ASIS is identified, the transducer is aligned with the pubic ramus and rotated at approximately 45 degrees, parallel to the inguinal crease. The transducer then slides medially along this axis until the anterior inferior iliac spine (AIIS), iliopubic eminence (IPE), and the psoas tendon is clearly identified, serving as anatomic landmarks. Sliding the probe distally or gently tilting the caudal will expose the head of the femur. Returning to the initial starting position, a standard 22 gauge spinal needle is inserted in-plane, from lateral to medial, in the plane between the psoas tendon and the pubic ramus. 20 ml 0.25% bupivacaine diluted with preservative free normal saline then deposited in this plane, lifting the psoas tendon. Care should be taken to avoid puncturing the psoas tendon.
  Arms: PENG Group

SUMMARY:
To study the efficacy of the PENG block on the duration of postoperative analgesia. There are two groups of patients, who are undergoing hip joint surgeries, one group (Control Group) will receive spinal anesthesia only while the other group (PENG Group) will receive PENG block before spinal anesthesia.

DETAILED DESCRIPTION:
Research Question:

Is PENG block effective in prolonging the duration of postoperative analgesia when compared to patients undergoing spinal anesthesia only?

Research Hypothesis:

PENG block is effective in prolonging the duration of postoperative analgesia and reducing postoperative pain.

Aim:

To improve the outcome of hip joint surgeries by decreasing the postoperative pain and early mobilization by performing PENG block to patients undergoing hip joint surgeries.

Method of randomization:

This clinical trial will be randomized through computer software that generates random number table and patients will be allocated randomly to one of the two groups.

Sample size:

The sample size was determined by using the following equation:(Charan J et al. 2013) N =(2 δ^(2 ) 〖(Z_α+ Z_β)〗^2)/D^2 δ=Standard deviation of the outcome = 6.7 (Pascarella et al., 2021). Z_α= The value for a type I error of 5% = 1.96 Z_β=The value for a type II error of 20% = 0.84 D^2= The effect size = 36 (Pascarella et al., 2021).

By calculation:

N = 19 per group. So, the total sample size is 38.

Procedures:

After getting the informed consent from the patient, the patient will be allocated into one of the study groups according to randomization.

ASA standard monitors will be attached to the patient, a wide pore cannula (18G) will be inserted then a premedication with 50 -100 mcg of fentanyl and 1-2 mg midazolam intravenously will be given.

PENG group: PENG block will done under complete aseptic condition with 20 ml 0.25% bupivacaine diluted with normal saline Control group: no block will be done. Both groups will be anesthetized using spinal anesthesia with Bupivacaine

Study Variables:

Independent variables: age, sex, weight, height, body mass index (BMI), elective or emergency surgery, duration of surgery, American Society of Anesthesiologists physical status classification (ASA score), occupation, fracture site, type of trauma, timing (operating room entry- PENG block time- start of spinal anesthesia- start of surgery- end of surgery ).

Dependent variables: Postoperative pain, adverse events, and postoperative motor assessment, hemodynamics, the first request of analgesia & total analgesia required, adverse events such as nausea vomiting & sedation, pain scores at preparation room, after PENG block, during sitting for spinal anesthesia, at end of the surgery, postoperative intervals(rest & movement).

ELIGIBILITY:
Inclusion Criteria:

* Patients with hip fracture who will be subjected to surgical treatment
* ASA physical status 1, 2

Exclusion Criteria:

* Patients with chronic pain before surgery (taking opioids).
* Patients with multiple trauma
* Patients who could not assess pain reliably (dementia).
* Substance abuse and prolonged intake of sedative drugs.
* Morbid obese patients (BMI>35).
* Patients who have open wounds or infection at the site of the block.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
The time of first request of analgesia in both groups | 24 hours postoperative
  The time of first request of analgesia in both groups in minutes

SECONDARY OUTCOMES:
Evaluate the morphine consumption over the first 24 hours. | 24 hours postoperative
  total dose of morphine in the first hours after surgery
Evaluate the regaining of motor function of quadriceps muscle in both groups | 24 hours postoperative
  Evaluate the motor function of quadriceps muscle by Medical research council (MRC) scale
The incidence of occurrence of side effects related to the technique and medications in both groups | 24 hours postoperative
  Nausea, vomiting
difference in Visual Analogue Score (VAS) pain score in the first 24 hours postoperative between the two groups | first 24 hours postoperative
  VAS pain score from 0-10 while 0 means no pain and 10 means the worst pain, at preparation room, after PENG block, during sitting for spinal anesthesia, at end of surgery, postoperative intervals(rest & movement).

CONTACTS AND LOCATIONS:
Locations (1):
- Suez Canal University, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR